CLINICAL TRIAL: NCT05896371
Title: PROstate-specific Membrane Antigen DosImetry-Guided EndoradiotherapY: a Phase 1/2 Study of Personalized PSMA Radiopharmaceutical Therapy (PRODIGY-1)
Brief Title: A Phase 1/2 Study of Personalized PSMA Radiopharmaceutical Therapy
Acronym: PRODIGY-1
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-6822
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Prostate Cancer; Metastatic Cancer; Metastatic Prostate Cancer
Keywords: Prostate-Specific Membrane Antigen; 177Lu-PSMA; Radiopharmaceutical Therapy; Dosimetry; Personalized
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A (Experimental): Lower risk of toxicity (no risk factor)
  Interventions: Drug: 177Lu-PSMA-I&T - escalating renal absorbed dose; Drug: 177Lu-PSMA-I&T - recommended phase 2 regime
- Cohort B (Experimental): Extensive bone metastasis
  Interventions: Drug: 177Lu-PSMA-I&T - escalating renal absorbed dose; Drug: 177Lu-PSMA-I&T - recommended phase 2 regime
- Cohort C (Experimental): Decreased bone marrow reserve
  Interventions: Drug: 177Lu-PSMA-I&T - escalating renal absorbed dose; Drug: 177Lu-PSMA-I&T - recommended phase 2 regime
- Cohort D (Experimental): Renal function impairment
  Interventions: Drug: 177Lu-PSMA-I&T - escalating renal absorbed dose; Drug: 177Lu-PSMA-I&T - recommended phase 2 regime
- Cohort E (Experimental): Higher risk of toxicity (more than one risk factor and others)
  Interventions: Drug: 177Lu-PSMA-I&T - escalating renal absorbed dose; Drug: 177Lu-PSMA-I&T - recommended phase 2 regime

INTERVENTIONS:
Drug: 177Lu-PSMA-I&T - escalating renal absorbed dose — Personalized 177Lu-PSMA-I&T injected activity
Drug: 177Lu-PSMA-I&T - recommended phase 2 regime — Personalized 177Lu-PSMA-I&T injected activity

SUMMARY:
The goal of this clinical trial is to study a personalized regime of lutetium-177 (177Lu) prostate-specific membrane antigen (PSMA) radiopharmaceutical therapy (RPT) in patients with progressive and/or symptomatic, inoperable PSMA-expressing cancers of prostatic or other origins.

The main questions it aims to answer are:

* To establish a dosimetry-based, personalized regime of 177Lu-PSMA
* To report on the efficacy of personalized 177Lu-PSMA

Participants (stratified by risk factors of toxicity) will receive up to 6 cycles of a personalized activity of 177Lu-PSMA based on renal dosimetry. In the phase 1, the prescribed absorbed dose to the kidney will be escalated, to determine the regime that will be administered in the phase 2. The best response within 12 months after the first cycle will be assessed. Salvage treatment of 3 cycles may be offered to responders after re-progression.

ELIGIBILITY:
Inclusion Criteria:

* >18 y.o. adults able to provide consent
* Inoperable or metastatic PSMA-expressing cancer, with significant PSMA expression defined as uptake in at least one lesion that is superior to that of the liver on PSMA positron-emission tomography (PET) within 3 months prior to enrolment
* Cancer progression documented within 3 months prior to enrolment as per the investigator's assessment, without initiation of another anti-cancer treatment since (excluding palliative radiation therapy to a minority of the tumor burden), unless that anti-cancer treatment was stopped prematurely because of intolerance
* For participants with a cancer other than mCRPC, a recommendation from a multidisciplinary tumor board (MDT) in favor of PSMA RPT must be obtained

Exclusion Criteria:

* Platelets < 50 x 106/L
* Absolute neutrophil count (ANC) < 1.0 x 106/L
* Eastern Cooperative Oncology Group (ECOG) 4 or prognosis < 3 months, for cancer-related or other serious medical conditions, as per investigator's assessment
* Known presence of central nervous system metastasis at risk of complication, which cannot be adequately stabilized (e.g. radiotherapy or corticoid prophylaxis), as per investigator's assessment
* Any condition that would limit the ability to comply with the study protocol, as per investigator's assessment
* Pregnancy or breastfeeding (e.g. for female participants with non-prostate cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2028-03 (Estimated); Primary Completion 2033-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of dose-limiting toxicities (DLTs) | 12 weeks
Phase 2: Overall response rate (ORR) | Up to 12 months
Phase 2: Biochemical response rate (PSA50) | Up to 12 months

SECONDARY OUTCOMES:
Frequency and grades of treatment-related adverse events (AEs) | Up to 12 months
Delayed AEs of particular interest | Up to 5 years
Phase 1: Overall response rate (ORR) | Up to 12 months
Phase 1: Biochemical response rate (PSA50) | Up to 12 months
Quality of life patient-reported outcome measures (PROMs) response rates | Up to 12 months
Progression-free survival (PFS) | Up to 5 years
Overall survival (OS) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Mathieu Beauregard, MD,MSc,FRCPC, Principal Investigator — CHU de Québec - Université Laval